CLINICAL TRIAL: NCT02313532
Title: Treatment of Febrile Infectious Disease Among Children in Hadera District Given the Final Diagnosis. Descriptive Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0092-14-HYMC
Record Dates: First submitted 2014-12-07; First posted 2014-12-10 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Febrile Illness Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Study goal - to describe pediatric patients with febrile disease that administered to the emergency department (ED) of hillel-yaffe hospital, according to arrival diagnosis, ED diagnosis, given therapy, and therapy concordance with the guidelines and final diagnosis.

This research will describe cases that arrived to the hospital with acute febrile disease (up to seven days of fever), the antibiotic treatment given in the community according to the anamnesis and the community physician letter, therapy concordance with the guidelines, the ED diagnosis and changes in therapy, and final diagnosis according to extended microbiological examinations and panel of infectious disease specialists.

DETAILED DESCRIPTION:
Major goal:

To describe cases that arrived to the pediatric ED with acute febrile illness (up to 7 days of fever) and the final diagnosis they received. To describe the antibiotic treatment given in the community as described in the anamnesis and referral letter, the concordance of the treatment to the therapeutic guidelines, the diagnosis given in the ED and the change in Antibiotic treatment, and the final diagnosis given after extended microbiologic tests were taken from a panel of infectious diseases specialists.

Minor goals:

1. Describing cohort of pediatric patients with acute febrile illness according to anamnesis, physical examination as a clarifying value to the final diagnosis.
2. Describing the antibiotic treatment given in the community and its concordance with therapeutic guidelines.
3. Describing patients referred to the ED after beginning antibiotic treatment
4. Describing patients arrived with sore throat that a diagnostic test for GAS was taken before antibiotic treatment was started.
5. Describing the difference between the antibiotic treatment given at the community, the treatment given at the hospital and the concordance to therapeutic guidelines
6. Describing the concordance between community diagnosis, in hospital diagnosis and the final diagnosis

Study assumption:

To create a map of infectious agents for children presenting with febrile illness, to decide which antibiotic prescribed was correct according to the final diagnosis. We assume that many of the given antibiotic treatments were incorrect to the final diagnosis.

Methodology:

Background:

Ruling out diagnosis of acute febrile illness in the ED is usually done relying on history, physical examination, routine laboratory tests (complete blood count, CRP, pro-calcitonin, urine dipstick), cultures (blood, urine. CSF, stool, throat culture etc.), imaging studies (Chest X-ray, ultra-sonography etc.) and other tests (lumbar puncture, serology, PCR etc.). the study:" Validation of markers for diagnosing the source of infection in pediatric febrile patient" number 0071-10-HYMC ("curiosity" study, see appendix A) is a prospective trial started in 2010 set in Hillel-yaffe hospital in Hadera, Israel. In this study patients with up to seven days of febrile illness, are recruited from the ED or pediatric department, history is taken that includes the home given therapy, blood tests are taken for complete blood count (CBC), culture and C-reactive peptide (CRP), imaging examinations are taken according to each case, PCR and Serology tests are taken to discern between number of agents (appendix A) and the final diagnosis is decided by a panel of infectious diseases specialists.

Research Method

Using "curiosity" study database for patients that recruited from the ED or pediatric department in Hillel-yaffe hospital. Usage of database will give the next data:

1. Final diagnosis of all patients, dividing the diagnosis for viral and bacterial and type of pathogen
2. Referral diagnosis, ED diagnosis, pediatric department diagnosis in concordance of the final diagnosis
3. The antibiotic treatment according to the referral letter and history and its concordance with therapeutic guidelines.
4. Changes or decision to stop antibiotic treatment in the hospital
5. Weather antibiotic therapy started at the community might interfere with making the right diagnosis (for example - antibiotic treatment started before urine culture was taken, GAS culture and rapid test taken)

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 7 days to 18 years.
2. Body temperature that is higher than 37.5°C (Rectal or Oral).
3. Informed consent obtained from parents.

Exclusion Criteria:

1. Children with fever that is longer than 7 days.
2. Children diagnosed with immunodeficiency.
3. Children that receive chemotherapy.
4. Children treated with high dose steroids.

Ages: 7 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Research population A sum of 500 patients recruited to the "curiosity" study in Hillel-yaffe hospital
  Inclusion criteria:
  1. Children aged 7 days to 18 years.
  2. Body temperature that is higher than 37.5°C (Rectal or Oral).
  3. Informed consent obtained from parents.
  Exclusion criteria:
  1. Children with fever that is longer than 7 days.
  2. Children diagnosed with immunodeficiency.
  3. Children that receive chemotherapy.
  4. Children treated with high dose steroids.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
pathogen map of febrile illness | 1 year

SECONDARY OUTCOMES:
antibiotic over use map | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: or kriger, m.d, Study Director — study coordinator
Locations (1):
- Hillel Yaffe MC,, Hadera, Israel

REFERENCES:
- [Background] Bergus GR, Levy BT, Levy SM, Slager SL, Kiritsy MC. Antibiotic use during the first 200 days of life. Arch Fam Med. 1996 Oct;5(9):523-6. doi: 10.1001/archfami.5.9.523. PMID 8930223
- [Background] Scheifele D, Halperin S, Pelletier L, Talbot J. Invasive pneumococcal infections in Canadian children, 1991-1998: implications for new vaccination strategies. Canadian Paediatric Society/Laboratory Centre for Disease Control Immunization Monitoring Program, Active (IMPACT). Clin Infect Dis. 2000 Jul;31(1):58-64. doi: 10.1086/313923. Epub 2000 Jul 24. PMID 10913397
- [Background] Whitney CG, Farley MM, Hadler J, Harrison LH, Lexau C, Reingold A, Lefkowitz L, Cieslak PR, Cetron M, Zell ER, Jorgensen JH, Schuchat A; Active Bacterial Core Surveillance Program of the Emerging Infections Program Network. Increasing prevalence of multidrug-resistant Streptococcus pneumoniae in the United States. N Engl J Med. 2000 Dec 28;343(26):1917-24. doi: 10.1056/NEJM200012283432603. PMID 11136262
- [Background] Seppala H, Nissinen A, Jarvinen H, Huovinen S, Henriksson T, Herva E, Holm SE, Jahkola M, Katila ML, Klaukka T, et al. Resistance to erythromycin in group A streptococci. N Engl J Med. 1992 Jan 30;326(5):292-7. doi: 10.1056/NEJM199201303260503. PMID 1728733
- [Background] Ladhani S, Gransden W. Increasing antibiotic resistance among urinary tract isolates. Arch Dis Child. 2003 May;88(5):444-5. doi: 10.1136/adc.88.5.444. PMID 12716722
- [Background] Dagan R, Leibovitz E, Greenberg D, Yagupsky P, Fliss DM, Leiberman A. Dynamics of pneumococcal nasopharyngeal colonization during the first days of antibiotic treatment in pediatric patients. Pediatr Infect Dis J. 1998 Oct;17(10):880-5. doi: 10.1097/00006454-199810000-00006. PMID 9802628